CLINICAL TRIAL: NCT03598907
Title: Point-of-care (POC) Approach to Management of Coagulopathy in Lung Transplantation Versus Standard Approach and Their Effect on Primary Graft Dysfunction (PGD), Randomized Controlled Study
Brief Title: Point-of-care Management of Coagulopathy in Lung Transplantation
Status: Terminated | Type: Observational
Why Stopped: After interim statistical analysis, the study was preliminary stopped as data was in favour of POC approach. See tables of results.
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., associate professor, University Hospital, Motol
Other Study IDs: NV19-06-00471
Record Dates: First submitted 2018-06-30; First posted 2018-07-26 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplantation
Keywords: point of care; coagulopathy; lung transplantation; primary graft dysfunction
MeSH Terms: conditions — Hemostatic Disorders; Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard management of coagulopathy: The first group of existing ,,standard care" - the approach to bleeding patient will be based on clinical experience of the anaesthetist, practically meaning administering crystalloids, colloids (hydroxyethyl starch or gelatin), fresh frozen plasma and erythrocytes to restore normovolemia and platelets, fibrinogen, prothrombin complex concentrate, von Willebrand factor, tranexamic acid, all products giving ,,blindly" when it comes to diagnosis and treatment of coagulopathy.
  Interventions: Other: Fresh frozen plasma
- POC management of coagulopathy: group of ,,point-of-care" approach to the diagnosis and treatment of perioperative bleeding and coagulopathy will be conducted on the basis of the results of the POC methods ROTEM, PFA 200 and Multiplate (prothrombin complex concentrate, fibrinogen, platelets, von Willebrand factor, tranexamic acid). A solution of 5% albumin and erythrocytes (to keep haemoglobin level over 100 g/l as it is critical for normal primary haemostasis) will be used to keep normal circulating volume and to compensate for perioperative blood loss.

INTERVENTIONS:
Other: Fresh frozen plasma — Fresh frozen plasma will be used according to anaesthetist ,,blind,, decision
  Groups: Standard management of coagulopathy

SUMMARY:
Pulmonary transplantation is a very demanding surgical procedure, often accompanied by coagulopathy and severe perioperative bleeding. The most common complication that develops within the first 72 hours after surgery is primary graft dysfunction (PGD), up to 30% in the most severe form. The etiology of PGD is multifactorial. One of the causes may be the amount of perioperative blood loss. Intravascular volume is normally maintained by the administration of crystalloid and colloid solutions and fresh frozen plasma, which is also used to treat coagulopathy, however it is administered at the discretion of the anaesthetist and his experience, practically meaning ,,blindly". In the field of the allogeneous ischemic organ, these substitution solutions essentially become another allogeneous material and can cause undesired immunomodulation and contribute to the development of PGD. In our prospective randomized trial (120 patients), two patient groups will be investigated. In the first group, the coagulopathy and perioperative blood loss will be treated by the current standard approach, by ,,blind" administration of fresh frozen plasma, crystalloids and colloids. In the second group, the cause of coagulopathy will be diagnosed and treated according to the point-of-care (POC) results of ROTEM, PFA 200 and Multiplate. A colloidal solution of 5% albumin will be used to replace the circulating volume and maintain the oncotic pressure. Investigators assume that the POC management of coagulopathy and bleeding in the second group will lead to a reduction in perioperative bleeding, to reduced administration of infusion solutions, and thus to a reduction of the incidence of PGD.

DETAILED DESCRIPTION:
Introduction and project description:

Primary graft dysfunction (PGD) in lung transplant patients is described as acute pulmonary damage occurring early in lung transplantation (in the first 72 hours) (1, 2), sometimes referred to as ischemia - reperfusion injury (1). It is characterized by non-cardiac pulmonary edema and diffuse alveolar damage. Clinically, it is manifested by varying degrees of hypoxemia, along with diffuse infiltrates in the X-ray of the lung. There are more theories that try to explain the cause of PGD. A number of factors such as cold organ ischemia, mechanical irritation during organ reperfusion, immunological, inflammatory, microbiological factors, and many others associated with lung transplantation (2, 3) may play a roll. Depending on the severity of the clinical symptoms and the severity of X-ray findings according to International Society of Heart and Lung Transplantation (ISHLT) there are three types of PGD. The incidence of PGD in its worst form (Grade 3) in early post-transplantation period is being reported to be present in up to 30% and between 10-25% within 24-72 hours after organ reperfusion. Lighter forms of PGD (1st and 2nd degree) occur much more frequently (2,3). Lung affected by PGD is characteristically edematous and the gas exchange is significantly impaired due to damage to the endothelial barrier integrity of the vessels and the epithelial barrier of the lung tissue. The presence of PGD significantly increases the morbidity and mortality of patients and significantly prolongs the time spent in invasive mechanical ventilation, generally prolongs the time spent in intensive care unit and is a significant risk factor for development of chronic rejection of the transplanted lung (2,3).

Lung transplantation is a demanding surgical procedure often associated with the development of coagulopathy and significant bleeding, especially when extracorporeal membrane oxygenation (ECMO) is used perioperatively, which is practically used in the most cases. Blood loss is replaced by the administration of crystalloid and colloid solutions in order to maintain normovolemia and by administering FFP, which is also used to treat coagulopathy, despite the fact that the International Normalized Ratio (INR) of blood plasma is 1.5-1.6. These preparations are administered according to the anesthesiologist's experience and practically ,,blindly". However, their administration in patient significantly immunocompromised may mean a risk of immunomodulation and thus a deterioration of PGD. In addition, the administration of blood plasma is generally associated with higher morbidity and mortality of patients (1).

On the other hand, point-of-care (POC) monitoring of the hemocoagulation state using rotational thromboelastometry (ROTEM) and subsequent targeted coagulopathy therapy during the perioperative period and traumatic life threatening bleeding resulted in decreased bleeding intensity and consumption of transfusion products and this approach led to a reduction in morbidity and mortality of these patients (2,3).

Also, methods for evaluating primary haemostasis such as PFA 200 (platelet function analyzer) and aggregometry-Multiplate can be used as POC methods in the operating room, especially for the diagnosis of coagulopathy accompanying the use of ECMO, especially for the diagnosis of von Willebrand's disease (PFA 200) or for the diagnosis of thrombocytopathy (Multiplate) (1-4).

All methods ROTEM, PFA 200 and Multiplate are used to predict bleeding in cardiac surgery and hepatic transplantation, and targeted therapy based on their results is associated with a reduction in blood transfusion (FFP, platelets, erythrocytes) administration, reduced bleeding and reduced morbidity and mortality (5-7).

Therefore, it can reasonably be assumed that a similar positive benefit of this POC approach can be expected even in patients undergoing lung transplantation.

In this prospective controlled randomized study of 120 lung transplant patients, investigators want to compare the incidence of PGD between a group of patients treated by standard ,,blind" approach and a ,,new" POC approach. Investigators assume that in a group where diagnosis and therapy of coagulopathy and bleeding will be managed based on the results of the ROTEM, PFA 200 and Multiplate tests, the clot strength will be increased and this will lead to reduced perioperative blood loss, reduced administration of infusion solutions and FFP and this will subsequently lead to reduced incidence of PGD.

Hypothesis:

Point-of-care approach to diagnosis of perioperative coagulopathy with ROTEM, PFA 200 and Multiplate and its subsequent aimed therapy will improve blood clot and thus will reduce blood loss, fluid infusion, blood transfusion and subsequently the incidence of PGD.

Methodology:

Patients undergoing bilateral lung transplantation (120 patients) will be randomized into 2 groups using computerised generator of random numbers. The study protocol will be registered in the Clinical Research Database and a clinical trial number (CTN) will be obtained and written informed consent will be obtained from patients before lung transplantation.

The first group of existing ,,standard care" - the approach to bleeding patient will be based on clinical experience of the anaesthetist, practically meaning administering crystalloids, colloids (hydroxyethyl starch or gelatin), fresh frozen plasma and erythrocytes to restore normovolemia and platelets, fibrinogen, prothrombin complex concentrate, von Willebrand factor, tranexamic acid, all products giving ,,blindly" when it comes to diagnosis and treatment of coagulopathy.

The second group of ,,point-of-care" approach to the diagnosis and treatment of perioperative bleeding and coagulopathy will be conducted on the basis of the results of the POC methods ROTEM, PFA 200 and Multiplate (prothrombin complex concentrate, fibrinogen, platelets, von Willebrand factor, tranexamic acid). A solution of 5% albumin and erythrocytes (to keep haemoglobin level over 100 g/l as it is critical for normal primary haemostasis) will be used to keep normal circulating volume and to compensate for perioperative blood loss.

Blood samples will obtained and analysed by ROTEM, PFA 200 and Multiplate, as well as the level and function of von Willebrand factor (multimers assay, ristocetin cofactor and collagen binding assay) will be performed in all patients:

1. before lung transplantation, upon patient arrival to hospital before surgery (as a control)
2. after lung transplantation, during admission of patient to postoperative intensive care unit
3. in the ,,POC" group also in the operating room (ROTEM, Multiplate and PFA 200) during surgery

The PGD score will be evaluated post-operatively and in the following way: severity of PGD is defined in four degrees and is evaluated using partial arterial oxygen pressure (PaO2) and inspired fraction of oxygen ratio (FiO2) ratio and simultaneously evaluating X-ray finding of the lungs as soon as possible after reperfusion (time 0) and after 48 and 72 hours after lung reperfusion.

* Grade 0 - PaO2/FiO2 ratio of any value but no pulmonary edema on chest X-ray
* Grade 1 - PaO2/FiO2 > 300 and presence of pulmonary edema on chest X-ray
* Grade 2 - PaO2/FiO2 200 - 300 and and presence of pulmonary edema on chest X-ray
* Grade 3 - PaO2/FiO2 < 200 and presence of pulmonary edema on chest X-ray or patients in need of postoperative ECMO support or nitric oxide therapy

To exclude the possible thrombotic complication of any of these approaches, each patient will be screened ultrasonographically for venous thrombosis 72 hours postoperatively (vena poplitea, vena femoralis, vena jugularis, and vena subclavia bilat) and thrombotic complications will compared between groups.

Also other parameters will be compared between groups:

* clot strength and whole coagulation profile before and after surgery using ROTEM, PFA 200 and Multiplate and evaluation of the functional level of von Willebrand factor. Correlation of coagulation profile with blood loss in the operating room and postoperative blood loss will be also assessed.
* amount of perioperative blood loss in the operating room at the end of surgery and 24 hours after surgery (blood loss will measured as amount of blood in the suction container in operating room and as amount of blood in the chest drain in ICU postoperatively)
* number of transfusion products administered in operating room and in postoperative ICU
* duration of invasive and noninvasive mechanical ventilation and time to extubation (hours), duration of stay in the postoperative ICU and overall in hospital before discharge home (days)
* morbidity of patients (SOFA score at 24, 48 and 72 hours after lung transplantation), morbidity and mortality among patients in 30, 90 and 365 days
* incidence of lung graft rejection during whole period of hospitalisation

Time schedule: 4 years During the 3-years period recruitment of patients will be done and in the 4-th year data will be analysed and published in valuable journals.

Investigators expect a lower consumption of blood transfusion products and infusion solutions in the POC group.

In case of lower PGD incidence in the POC group investigators expect shorter time of mechanical ventilation, a shorter period of hospitalization at the postoperative ICU and in the hospital overall and a lower incidence of pulmonary graft rejection.

Investigators expect lower morbidity and mortality of patients in the POC group.

Investigators also believe that the POC approach will reduce the total hospitalisation costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Indicated for bilateral lung transplantation with diagnosis of interstitial pulmonary fibrosis, cystic fibrosis, chronic obstructive pulmonary disease, exogenous allergic alveolitis

Exclusion Criteria:

* Patients requiring plasmapheresis before lung transplantation
* Patients waiting for lung transplantation on ECMO (ECMO used as bridging to surgery)
* Patients undergoing simultaneous lung and heart transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old who are indicated for bilateral lung transplantation with diagnosis of interstitial pulmonary fibrosis, cystic fibrosis, chronic obstructive pulmonary disease, exogenous allergic alveolitis.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Durila, assoc.prof., Principal Investigator — University Hospital, Motol
Locations (1):
- University Hospital Motol, Department of Anaesthesiology and Intensive Care, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snell GI, Yusen RD, Weill D, Strueber M, Garrity E, Reed A, Pelaez A, Whelan TP, Perch M, Bag R, Budev M, Corris PA, Crespo MM, Witt C, Cantu E, Christie JD. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction, part I: Definition and grading-A 2016 Consensus Group statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2017 Oct;36(10):1097-1103. doi: 10.1016/j.healun.2017.07.021. Epub 2017 Jul 26. No abstract available. PMID 28942784
- [Background] Diamond JM, Arcasoy S, Kennedy CC, Eberlein M, Singer JP, Patterson GM, Edelman JD, Dhillon G, Pena T, Kawut SM, Lee JC, Girgis R, Dark J, Thabut G. Report of the International Society for Heart and Lung Transplantation Working Group on Primary Lung Graft Dysfunction, part II: Epidemiology, risk factors, and outcomes-A 2016 Consensus Group statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2017 Oct;36(10):1104-1113. doi: 10.1016/j.healun.2017.07.020. Epub 2017 Jul 26. No abstract available. PMID 28802530
- [Background] Gelman AE, Fisher AJ, Huang HJ, Baz MA, Shaver CM, Egan TM, Mulligan MS. Report of the ISHLT Working Group on Primary Lung Graft Dysfunction Part III: Mechanisms: A 2016 Consensus Group Statement of the International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 2017 Oct;36(10):1114-1120. doi: 10.1016/j.healun.2017.07.014. Epub 2017 Jul 24. No abstract available. PMID 28818404
- [Background] Gorlinger K, Saner FH. Prophylactic plasma and platelet transfusion in the critically Ill patient: just useless and expensive or even harmful? BMC Anesthesiol. 2015 Jun 9;15:86. doi: 10.1186/s12871-015-0074-0. PMID 26054337
- [Background] Keene DD, Nordmann GR, Woolley T. Rotational thromboelastometry-guided trauma resuscitation. Curr Opin Crit Care. 2013 Dec;19(6):605-12. doi: 10.1097/MCC.0000000000000021. PMID 24240827
- [Background] Hagemo JS, Christiaans SC, Stanworth SJ, Brohi K, Johansson PI, Goslings JC, Naess PA, Gaarder C. Detection of acute traumatic coagulopathy and massive transfusion requirements by means of rotational thromboelastometry: an international prospective validation study. Crit Care. 2015 Mar 23;19(1):97. doi: 10.1186/s13054-015-0823-y. PMID 25888032
- [Background] Mutlak H, Reyher C, Meybohm P, Papadopoulos N, Hanke AA, Zacharowski K, Weber CF. Multiple electrode aggregometry for the assessment of acquired platelet dysfunctions during extracorporeal circulation. Thorac Cardiovasc Surg. 2015 Feb;63(1):21-7. doi: 10.1055/s-0034-1383817. Epub 2014 Aug 1. PMID 25083831
- [Background] Kalbhenn J, Schlagenhauf A, Rosenfelder S, Schmutz A, Zieger B. Acquired von Willebrand syndrome and impaired platelet function during venovenous extracorporeal membrane oxygenation: Rapid onset and fast recovery. J Heart Lung Transplant. 2018 Aug;37(8):985-991. doi: 10.1016/j.healun.2018.03.013. Epub 2018 Mar 17. PMID 29650295
- [Background] Bogdanic D, Karanovic N, Mratinovic-Mikulandra J, Paukovic-Sekulic B, Brnic D, Marinovic I, Nonkovic D, Bogdanic N. The Role of Platelet Function Analyzer Testing in Cardiac Surgery Transfusion Management. Transfus Med Hemother. 2017 Apr;44(2):106-113. doi: 10.1159/000452863. Epub 2017 Feb 1. PMID 28503127
- [Background] Ellis J, Valencia O, Crerar-Gilbert A, Phillips S, Meeran H, Sharma V. Point-of-care platelet function testing to predict blood loss after coronary artery bypass grafting surgery: a prospective observational pilot study. Perfusion. 2016 Nov;31(8):676-682. doi: 10.1177/0267659116656774. Epub 2016 Jul 10. PMID 27388540
- [Background] Deppe AC, Weber C, Zimmermann J, Kuhn EW, Slottosch I, Liakopoulos OJ, Choi YH, Wahlers T. Point-of-care thromboelastography/thromboelastometry-based coagulation management in cardiac surgery: a meta-analysis of 8332 patients. J Surg Res. 2016 Jun 15;203(2):424-33. doi: 10.1016/j.jss.2016.03.008. Epub 2016 Mar 26. PMID 27363652
- [Background] Pearse BL, Smith I, Faulke D, Wall D, Fraser JF, Ryan EG, Drake L, Rapchuk IL, Tesar P, Ziegenfuss M, Fung YL. Protocol guided bleeding management improves cardiac surgery patient outcomes. Vox Sang. 2015 Oct;109(3):267-79. doi: 10.1111/vox.12279. Epub 2015 Apr 30. PMID 25930098
- [Background] Leon-Justel A, Noval-Padillo JA, Alvarez-Rios AI, Mellado P, Gomez-Bravo MA, Alamo JM, Porras M, Barrero L, Hinojosa R, Carmona M, Vilches-Arenas A, Guerrero JM. Point-of-care haemostasis monitoring during liver transplantation reduces transfusion requirements and improves patient outcome. Clin Chim Acta. 2015 Jun 15;446:277-83. doi: 10.1016/j.cca.2015.04.022. Epub 2015 Apr 25. PMID 25916692
- [Result] Durila M, Vajter J, Garaj M, Pollert L, Berousek J, Vachtenheim J Jr, Vymazal T, Lischke R. Rotational thromboelastometry reduces blood loss and blood product usage after lung transplantation. J Heart Lung Transplant. 2021 Jul;40(7):631-641. doi: 10.1016/j.healun.2021.03.020. Epub 2021 Mar 29. PMID 33934981
- [Result] Vajter J, Vachtenheim J Jr, Prikrylova Z, Berousek J, Vymazal T, Lischke R, Martin AK, Durila M. Effect of targeted coagulopathy management and 5% albumin as volume replacement therapy during lung transplantation on allograft function: a secondary analysis of a randomized clinical trial. BMC Pulm Med. 2023 Mar 9;23(1):80. doi: 10.1186/s12890-023-02372-0. PMID 36894877
- [Derived] Durila M, Vajter J, Garaj M, Smetak T, Hedvicak P, Berousek J, Vymazal T. Acquired primary hemostasis pathology detected by platelet function analyzer 200 seen during extracorporeal membrane oxygenation is sufficient to prevent circuit thrombosis: A pilot study. J Heart Lung Transplant. 2020 Sep;39(9):980-982. doi: 10.1016/j.healun.2020.05.015. Epub 2020 Jun 11. No abstract available. PMID 32591313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After performing an interim statistical analysis of the results in approximatelly the middle of the study, the project was prematurely terminated as it would have been unethical to continue.
Pre-assignment Details: Total number of patients anticipated in the study was 120, meaning 60 patients in every group.
Period: Overall Study
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
Started | 50 | 50
Completed | 36 | 31
Not Completed | 14 | 19
Not completed — Physician Decision | 14 | 19

BASELINE CHARACTERISTICS:
Groups:
- "Non POC" Group: the management of perioperative bleeding and coagulopathy and the administration of RBC, FFP, and PLT was based on the clinical experience of the anesthesiologist
- "POC Group": the management of perioperative bleeding and coagulopathy based on results of POC method such as ROTEM
- Total: Total of all reporting groups
Arm/Group | "Non POC" Group | "POC Group" | Total
Number analyzed (Participants) | 36 | 31 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 31 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 45 (16) | 50.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 25 | 20 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 31 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 36 | 31 | 67

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Blood Loss
Description: Total estimated blood loss measured during the perioperative period of lung transplantation (including intraoperative and immediate postoperative period).
Time Frame: From the beginning of surgery to 24 hours postoperatively
Population: All randomized patients who underwent lung transplantation
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Non POC Group: Bleeding and coagulopathy was managed based on clinical approach of anesthesiologist.
- POC Group: Bleeding and coagulopathy was managed according to results of point of care tests ROTEM, PFA 200 and Multiplate.
Arm/Group | Non POC Group | POC Group
Number analyzed (Participants) | 36 | 31
mL | 1043 (547) | 682 (399)

2. Other Pre Specified Outcome: Primary Graft Dysfunction (PGD)
Description: PGD 0-1 and 2-3 differences between POC versus Non-POC group. Primary graft dysfunction (PGD) in lung transplant patients is described as acute pulmonary damage occurring early in lung transplantation.
  The severity of PGD is defined in four degrees and is evaluated using partial arterial oxygen pressure (PaO2) and inspired fraction of oxygen ratio (FiO2) ratio and simultaneously evaluating X-ray finding of the lungs after surgery.
  * Grade 0 - PaO2/FiO2 ratio of any value but no pulmonary edema on chest X-ray
  * Grade 1 - PaO2/FiO2 > 300 and presence of pulmonary edema on chest X-ray
  * Grade 2 - PaO2/FiO2 200 - 300 and and presence of pulmonary edema on chest X-ray
  * Grade 3 - PaO2/FiO2 < 200 and presence of pulmonary edema on chest X-ray or patients in need of postoperative ECMO support or nitric oxide therapy
Time Frame: After surgery at 0 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
Number analyzed (Participants) | 36 | 31
Participants
  PGD 0-1 | 22 | 24
  PGD 2-3 | 14 | 7

3. Other Pre Specified Outcome: Primary Graft Dysfunction (PGD)
Description: PGD 0-1 and 2-3 differences between POC versus Non-POC group PGD 0-1 and 2-3 differences between POC versus Non-POC group. Primary graft dysfunction (PGD) in lung transplant patients is described as acute pulmonary damage occurring early in lung transplantation.
  The severity of PGD is defined in four degrees and is evaluated using partial arterial oxygen pressure (PaO2) and inspired fraction of oxygen ratio (FiO2) ratio and simultaneously evaluating X-ray finding of the lungs after surgery.
  * Grade 0 - PaO2/FiO2 ratio of any value but no pulmonary edema on chest X-ray
  * Grade 1 - PaO2/FiO2 > 300 and presence of pulmonary edema on chest X-ray
  * Grade 2 - PaO2/FiO2 200 - 300 and and presence of pulmonary edema on chest X-ray
  * Grade 3 - PaO2/FiO2 < 200 and presence of pulmonary edema on chest X-ray or patients in need of postoperative ECMO support or nitric oxide therapy
Time Frame: After surgry at 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
Number analyzed (Participants) | 36 | 31
Participants
  PGD 0-1 | 28 | 28
  PGD 2-3 | 8 | 3

4. Other Pre Specified Outcome: Primary Graft Dysfunction (PGD)
Description: PGD 0-1 and 2-3 differences between POC versus Non-POC group. PGD 0-1 and 2-3 differences between POC versus Non-POC group. Primary graft dysfunction (PGD) in lung transplant patients is described as acute pulmonary damage occurring early in lung transplantation.
  The severity of PGD is defined in four degrees and is evaluated using partial arterial oxygen pressure (PaO2) and inspired fraction of oxygen ratio (FiO2) ratio and simultaneously evaluating X-ray finding of the lungs after surgery.
  * Grade 0 - PaO2/FiO2 ratio of any value but no pulmonary edema on chest X-ray
  * Grade 1 - PaO2/FiO2 > 300 and presence of pulmonary edema on chest X-ray
  * Grade 2 - PaO2/FiO2 200 - 300 and and presence of pulmonary edema on chest X-ray
  * Grade 3 - PaO2/FiO2 < 200 and presence of pulmonary edema on chest X-ray or patients in need of postoperative ECMO support or nitric oxide therapy
Time Frame: After surgry at 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
Number analyzed (Participants) | 36 | 31
Participants
  PGD 0-1 | 27 | 26
  PGD 2-3 | 9 | 5

5. Other Pre Specified Outcome: Primary Graft Dysfunction (PGD)
Description: as for outcome 4
Time Frame: After surgry at 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
Number analyzed (Participants) | 36 | 31
Participants
  PGD 0-1 | 27 | 30
  PGD 2-3 | 9 | 1

ADVERSE EVENTS:
Time Frame: 72 hours after surgery
Description: Adverse events "non-POC" group "POC" group Thrombotic complications (n) 0 0 Mortality (n) 0 0
Groups:
- POC Management of Coagulopathy: group of ,,point-of-care" approach to the diagnosis and treatment of perioperative bleeding and coagulopathy will be conducted on the basis of the results of the POC methods ROTEM (prothrombin complex concentrate, fibrinogen, platelets, von Willebrand factor, tranexamic acid). A solution of 5% albumin and erythrocytes (to keep haemoglobin level over 100 g/l as it is critical for normal primary haemostasis) will be used to keep normal circulating volume and to compensate for perioperative blood loss.
Arm/Group | Standard Management of Coagulopathy | POC Management of Coagulopathy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03598907/Prot_000.pdf
  • Informed Consent Form (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03598907/ICF_001.pdf